CLINICAL TRIAL: NCT02963610
Title: A Phase I Study of Lenalidomide Plus Pembrolizumab in Patients With Relapsed and/or Refractory Solid Tumors With Phase II Expansion in Non-small Cell Lung Cancer
Brief Title: Phase I/II Study of Lenalidomide Plus Pembrolizumab in Patients With Solid Tumors With Expansion in Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated prematurely due to funding/support being withdrawn by grantor
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH-088
Record Dates: First submitted 2016-11-09; First posted 2016-11-15 (Estimated); Results first posted 2021-12-30 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Relapsed or Refractory Solid Tumors; Nonsmall Cell Lung Cancer
MeSH Terms: conditions — Recurrence; Carcinoma, Non-Small-Cell Lung | interventions — Lenalidomide; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab, Lenalidomide (Experimental): Phase I The treatment will be given on a 21-day cycle, with a dose of pembrolizumab given on day1(IV) and doses of lenalidomide given on day 1-14 (orally). The dose of pembrolizumab will be fixed at 200 mg. The dose of lenalidomide will depend upon the patient cohort. Cohort 1 will receive 10mg, Cohort II will receive 15mg and cohort 3 will receive 20mg of lenalidomide.
  Phase II The treatment will be given on a 21-day cycle, with a dose of pembrolizumab given on day1(IV) and doses of lenalidomide given on day 1-14 (orally). The dose of pembrolizumab will be fixed at 200 mg. Maximum Tolerated Dose (MTD) of lenalidomide as determined by the Phase I study will be given in Phase II study.
  Interventions: Drug: Lenalidomide; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide is a thalidomide analogue with immunomodulatory, anti-angiogenic, and antineoplastic effects. It is administered as a pill taken orally. It has completed phase III study evaluation and has FDA indications for use in certain patients with multiple myeloma, myelodysplastic syndrome, and mantle cell lymphoma.
  Other Names: Revlimid
Drug: Pembrolizumab — Pembrolizumab is a humanized IgG4 monoclonal antibody which targets the PD-1 receptor, thus inhibiting the interaction between PD-1 and its ligands, PD-L1 and PD-L2 respectively. It is administered as an IV infusion. This drug has several studies in patients with solid tumors and currently has an FDA indication for use in patients with melanoma and non-small cell lung cancer.
  Other Names: Keytruda

SUMMARY:
For the phase I component of the trial a classic 3 + 3 dose escalation design will be utilized, with a fixed dose of pembrolizumab and an escalating dose of the lenalidomide. The patient population will all have histologically confirmed advanced solid tumor malignancy. The primary endpoint for the phase I component of this protocol will be determining the maximum tolerated dose (MTD) of lenalidomide in combination with pembrolizumab.

The phase II component of this trial will utilize a two stage design, initially enrolling 13 patients, followed by 13 more patients if the early stopping criteria are not met. The target population will include patients with histologically confirmed diagnoses of non-small cell lung carcinoma, regardless of histologic subtype; who have completed one line of standard therapy. The primary endpoint for the phase II component of this protocol will be determining efficacy as measured by progression free survival (PFS)

DETAILED DESCRIPTION:
Phase I The study will plan to enroll 3 patients in an initial cohort, to receive the dose level 1 of lenalidomide (10 mg PO) on days 1-14 of a 21-day cycle, and pembrolizumab (200 mg IV) on day 1. Patients will be evaluated for toxicities after initiation of treatment. If there are no DLTs for the initial 3 patients after one cycle, the next dosing cohort will open, with another 3 patients. Similarly, if the second cohort of patients receives the dose level 2 of lenalidomide (15 mg) for one cycle without DLT, then the third and final cohort will open. When the third cohort testing the dose level 3 of lenalidomide (20 mg) has completed one cycle, the phase I component of the trial will be completed. Standard phase I, 3 + 3 design rules will be utilized as follows: if 1 out of 3 patients experiences a DLT at certain dose level, then 3 more patients will be enrolled at the same level. If 2 out of 6 patients experience DLT at a certain dose level, 3 additional patients are added at the next lower level. Dose reduction is continued until at most 1 of 6 patients experiences DLT. The highest level with at most 1 of 6 patients DLT will be declared MTD. If no dose level achieves this criterion the trial will be discontinued for excess toxicity.

Phase II A pre-treatment (archival) and fresh tumor sample will be needed for participation in trial. PD-L1 expression levels in both samples will be determined to assess the role of chemotherapy on expression level and pattern of this biomarker. Baseline blood samples will be collected for immunologic correlates prior to treatment on Day 1 of Cycle 1 and post treatment at 2, 4, 24 hours. Samples will also be collected prior to treatment on Day 1 of Cycle 2, and at time of progression. Baseline CT scan of the chest and abdomens will be obtained within 30 days prior to the initiation of cycle 1. CT scan with contrast or MRI with contrast of the brain will also be obtained within 30 days prior to the initiation of cycle 1. Time to progression will be measured with disease imaging following every 2 cycles of therapy with a three-day window (+ or -). Patients will continue treatment until disease progression or unacceptable toxicity or two years of therapy. Overall survival will be assessed every 3 months during long term follow up

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologically or cytologically confirmed metastatic solid tumor malignancy for the phase I component. The phase II component will require patients to have histologically or cytologically confirmed non-small cell lung carcinoma regardless of histology.
2. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension in accordance with RECIST criteria v. 1.1.
3. For participation in the Phase II portion, patients must have completed at least one line of prior therapy. For participation in the Phase I portion, patients must have completed either one or two lines of prior therapy.
4. Treatment on this protocol may begin as long as the patient has recovered from toxicities of prior therapy at the discretion of the treating physician. Patients with NSCLC harboring an EGFR, ALK or ROS-1 alteration must have progressed through at least one prior therapy with appropriate molecularly targeted agents.
5. Age > 18 years.
6. ECOG performance status 0 or 1.
7. Patients must have normal organ and marrow function
8. Ability to understand and willingness to sign a written informed consent and HIPAA consent document.
9. Palliative radiation for treatment of painful bone metastasis, control of hemoptysis or treatment of small asymptomatic brain metastasis that become symptomatic during on protocol treatment is allowed. Protocol treatment will be delayed until recovery from radiation at the discretion of the treating physician.
10. A core tumor biopsy obtained after progression on the last treatment must be available at study entry for the phase II portion of the study. Any available archival tissue (for both phase I and II) will also be collected.
11. Female subject of childbearing potential must have a negative serum pregnancy 10-14 days prior to registration, and again within 24 hours prior to the first dose of Lenalidomide,.
12. Female subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication.
13. Male subjects of childbearing potential must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
14. Ten patients with a diagnosis of NSCLC who have disease progression per investigator's assessment who are on anti PD-1 or PD-L1 therapies will be allowed to enroll in the phase II part of this study but must be switched to treatment per this protocol.

Exclusion Criteria:

1. Patients who have had chemotherapy or radiotherapy within14 days prior to entering the study. Patients may not be currently receiving any other investigational agents or immunomodulatory agents (e.g. ipilimumab). Patients treated with prior PD-1 or PD-L1 directed therapies are ineligible for the phase I portion.
2. Patients who, at the discretion of the treating physician, have not recovered from adverse events due to agents administered earlier.
3. Patients with active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
4. Patients with untreated symptomatic brain metastases. Patients with treated brain metastases will be allowed if brain imaging obtained within 30 days of trial enrollment reveals stable disease. Patients with small asymptomatic brain metastasis are allowed to enroll. Patients on steroids doses higher than 10 mg of prednisone (or its equivalent) are excluded.
5. Patients with interstitial lung disease or active, noninfectious pneumonitis.
6. Patient who have received a live vaccine within 30 days prior to Cycle 1 Day 1.
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (including HIV, hepatitis B, hepatitis C), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, cirrhosis, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Patients with known hypersensitivity to thalidomide or lenalidomide or pomalidomide.
9. Patients with peripheral neuropathy of grade ≥3. Patients with painful grade 2 neuropathy are also excluded.
10. Pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2017-10-03 (Actual); Study Completion 2018-03-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab, Lenalidomide: Phase I The treatment will be given on a 21-day cycle, with a dose of pembrolizumab given on day1(IV) and doses of lenalidomide given on day 1-14 (orally). The dose of pembrolizumab will be fixed at 200 mg. The dose of lenalidomide will depend upon the patient cohort. Cohort 1 will receive 10mg, Cohort II will receive 15mg and cohort 3 will receive 20mg of lenalidomide.
  Phase II The treatment will be given on a 21-day cycle, with a dose of pembrolizumab given on day1(IV) and doses of lenalidomide given on day 1-14 (orally). The dose of pembrolizumab will be fixed at 200 mg. Maximum Tolerated Dose (MTD) of lenalidomide as determined by the Phase I study will be given in Phase II study.
  Lenalidomide: Lenalidomide is a thalidomide analogue with immunomodulatory, anti-angiogenic, and antineoplastic effects. It is administered as a pill taken orally. It has completed phase III study evaluation and has FDA indications for use in certain patients with multiple myeloma, myelodysplastic syndrome, and mantle cell lymphoma.
  Pembrolizumab: Pembrolizumab is a humanized IgG4 monoclonal antibody which targets the PD-1 receptor, thus inhibiting the interaction between PD-1 and its ligands, PD-L1 and PD-L2 respectively. It is administered as an IV infusion. This drug has several studies in patients with solid tumors and currently has an FDA indication for use in patients with melanoma and non-small cell lung cancer.
Period: Overall Study
Arm/Group | Pembrolizumab, Lenalidomide
Started | 3
Completed | 0
Not Completed | 3
Not completed — Study terminated prematurely due to funding/support being withdrawn by grantor. No analyses occurred | 3

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab, Lenalidomide
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 2
  Black or African American | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Maximum Tolerated Dose (MTD) of Lenalidomide in Combination With a Fixed Dose of Pembrolizumab in Subjects With Relapsed and/or Refractory Solid Tumors.
Description: Maximum tolerated dose of Lenalidomide
Time Frame: Day 22 of cycle 1
Population: Study terminated prematurely due to funding/support being withdrawn by grantor. No analyses occurred
Groups:
- Experimental: Pembrolizumab, Lenalidomide: Phase I The treatment will be given on a 21-day cycle, with a dose of pembrolizumab given on day1(IV) and doses of lenalidomide given on day 1-14 (orally). The dose of pembrolizumab will be fixed at 200 mg. The dose of lenalidomide will depend upon the patient cohort. Cohort 1 will receive 10mg, Cohort II will receive 15mg and cohort 3 will receive 20mg of lenalidomide.
  Phase II The treatment will be given on a 21-day cycle, with a dose of pembrolizumab given on day1(IV) and doses of lenalidomide given on day 1-14 (orally). The dose of pembrolizumab will be fixed at 200 mg. Maximum Tolerated Dose (MTD) of lenalidomide as determined by the Phase I study will be given in Phase II study.
  Lenalidomide: Lenalidomide is a thalidomide analogue with immunomodulatory, anti-angiogenic, and antineoplastic effects. It is administered as a pill taken orally. It has completed phase III study evaluation and has FDA indications for use in certain patients with multiple myeloma, myelodysplastic syndrome, and mantle cell lymphoma.
  Pembrolizumab: Pembrolizumab is a humanized IgG4 monoclonal antibody which targets the PD-1 receptor, thus inhibiting the interaction between PD-1 and its ligands, PD-L1 and PD-L2 respectively. It is administered as an IV infusion. This drug has several studies in patients with solid tumors and currently has an FDA indication for use in patients with melanoma and non-small cell lung cancer.
Arm/Group | Experimental: Pembrolizumab, Lenalidomide
Number analyzed (Participants) | 0

2. Primary Outcome: To Determine Efficacy as Measured by Progression Free Survival (PFS) in Non-small Cell Lung Cancer Patients
Description: PFS
Time Frame: up to 3 years
Population: Study terminated prematurely due to funding/support being withdrawn by grantor. No analyses occurred
Arm/Group | Pembrolizumab, Lenalidomide
Number analyzed (Participants) | 0

3. Secondary Outcome: Assess Antitumor Activity of the Combination as Measured by Objective Response Rate (ORR)
Description: ORR
Time Frame: upto 2 years
Population: Study terminated prematurely due to funding/support being withdrawn by grantor. No analyses occurred
Arm/Group | Pembrolizumab, Lenalidomide
Number analyzed (Participants) | 0

4. Secondary Outcome: Assessment of PD-L1 Expression by Immunohistochemistry
Description: PD-1 expression will be used to correlate with the treatment response
Time Frame: upto 2 years
Population: Study terminated prematurely due to funding/support being withdrawn by grantor. No analyses occurred
Arm/Group | Pembrolizumab, Lenalidomide
Number analyzed (Participants) | 0

5. Secondary Outcome: Proportions of Blood Immune Cells by Flow Cytometry
Description: Amount of CD45, CD3, CD4, CD8 (T cells), CD19 (B cells), CD14, CD16 (monocytes), CD56 (NK cells), CD11c, HLA-DR, CD303, CD66b (myeloid - DCs and granulocytes).
Time Frame: upto 2 years
Population: Study terminated prematurely due to funding/support being withdrawn by grantor. No analyses occurred
Arm/Group | Pembrolizumab, Lenalidomide
Number analyzed (Participants) | 0

6. Secondary Outcome: Assesment of Cytokine Profiles Using Luminex
Description: Th1/Tc1 responses ( IFN-g, TNF, IL-2), Th2/Tc1 responses (IL-4, IL-5, IL-10), pro-inflammatory innate responses (IFN-α, IL-1β, IL-6, IL-17), homeostatic lymphocyte expansion (IL-7, IL-15), and chemotaxis of immune cells (IP-10, MCP-1, MIP-1α, MIP-1β, RANTES) will be measured
Time Frame: upto 2 years
Population: Study terminated prematurely due to funding/support being withdrawn by grantor. No analyses occurred
Arm/Group | Pembrolizumab, Lenalidomide
Number analyzed (Participants) | 0

7. Secondary Outcome: Determine Specific NK Cell Responses by NK Degranulation Assay by Flow Cytometry
Description: CD107A expression after 2 hour co-culture with the EBV-transformed B cell line, 721.221, without and with rituximab (ADCC conditions).
Time Frame: upto 2 years
Population: Study terminated prematurely due to funding/support being withdrawn by grantor. No analyses occurred
Arm/Group | Pembrolizumab, Lenalidomide
Number analyzed (Participants) | 0

8. Secondary Outcome: Assessment of Activation Markers on Immune Cells by Flow Cytometry
Description: Activation markers will include CD69, CD25, HLA-DR, IL-15Ra, perforin, Ki67, NKp44, CD57
Time Frame: upto 2 years
Population: Study terminated prematurely due to funding/support being withdrawn by grantor. No analyses occurred
Arm/Group | Pembrolizumab, Lenalidomide
Number analyzed (Participants) | 0

9. Secondary Outcome: Determine Immune Composition of Tumors Using PanCancer Immune Profiling Panel by Nanostring Technology
Description: Expression of genes involved in immune responses
Time Frame: upto 2 years
Population: Study terminated prematurely due to funding/support being withdrawn by grantor. No analyses occurred
Arm/Group | Pembrolizumab, Lenalidomide
Number analyzed (Participants) | 0

10. Secondary Outcome: From Patients That Were Previously Treated With an Anti-PD1 Antibody, we Will Determine Resistance Overcome Due to the Treatment With Combination Assessed by Overall Response Rate.
Description: number of patients that overcome the resistance of previous anti-pD-1 therapy
Time Frame: upto 2 years
Population: Study terminated prematurely due to funding/support being withdrawn by grantor. No analyses occurred
Arm/Group | Pembrolizumab, Lenalidomide
Number analyzed (Participants) | 0

11. Secondary Outcome: Determine Specific T Cell Responses by Determining Differentiation Status of T Cells by Flow Cytometry
Description: Differentiation status of CD4 and CD8 T cells (naïve/effector memory/central memory/regulatory/delta-gamma TCR) as defined by: CD62L, CD45RA, CD127, CD25.
Time Frame: upto 2 years
Population: Study terminated prematurely due to funding/support being withdrawn by grantor. No analyses occurred
Arm/Group | Pembrolizumab, Lenalidomide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Pembrolizumab, Lenalidomide
All-Cause Mortality (participants affected / at risk) | 2/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab, Lenalidomide (N=3)
Constipation (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Fecal incontinence (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Hypoalkemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 2
Hypothyroidism (Endocrine disorders) | 1
Photophobia (Eye disorders) | 1
Watering eyes (Eye disorders) | 1
Chills (General disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 1
Weight loss (Investigations) | 1
Dizziness (Nervous system disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-09): https://cdn.clinicaltrials.gov/large-docs/10/NCT02963610/Prot_SAP_000.pdf